CLINICAL TRIAL: NCT00761592
Title: Comparison of Two Botulinum Type A Products in the Treatment of Blepharospasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALLBL001
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: Botulinum Toxin Type A 900kDa
- 2 (Active Comparator)
  Interventions: Biological: Botulinum Toxin Type A 150kDa

INTERVENTIONS:
Biological: Botulinum Toxin Type A 900kDa — 6 to 16 injections, with maximum of 21, at a dose of ≥20U/eye (≥40U total dose)
  Other Names: BOTOX®
  Arms: 1
Biological: Botulinum Toxin Type A 150kDa — 6 to 16 injections, with a maximum of 21, at a dose of ≥20U/eye (≥40U total dose)
  Other Names: Xeomin®
  Arms: 2

SUMMARY:
This pilot study estimates the treatment effects of two different types of botulinum toxin type A in the treatment of Blepharospasm. Blepharospasm is characterised by excessive contraction of the muscles around the eye and can lead to repetitive blinking or sustained closure of the eyelids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with benign essential blepharospasm
* Received ≥20U/eye of BOTOX® for at least one visit prior to study entry and required, in the investigators opinion, the same dose at the study injection visit.
* Combined Jankovic Rating Score of >2

Exclusion Criteria:

* Female subjects who were pregnant, breastfeeding, or who were of childbirth potential and not practicing birth control.
* Profound atrophy of the muscles in the target area(s) of injection.
* Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
* Known significantly impaired renal and/or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Germany (3):
  - Bonn
  - Wiesbaden
  - Zwickau

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Started | 32 | 33
Completed | 31 | 32
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa | Total
Number analyzed (Participants) | 31 | 33 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 70.7 (10.7) | 67.1 (12.1) | 68.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — One patient from group 1 withdrew consent after first injection, thus efficacy data was not gathered for this patient
  Participants
    Female | 20 | 19 | 39
    Male | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Blepharospasm Disability Index
Description: Blepharospasm Disability Index is a validated 5-point scale (0-4) with six items (e.g., reading, driving a vehicle).
  0 - no impairment, 1 - mild impairment, 2 - moderate impairment, 3 - severe impairment, 4 - not possible due to disease, N/A - Not applicable.
  The total score ranged from 0 (no impairment) to 24 (not possible due to disease). A negative change from baseline indicated improvement.
Time Frame: Baseline to Week 4
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: Points on Scale
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Number analyzed (Participants) | 31 | 33
Points on Scale | -2.8 (5.3) | -1.3 (3.7)

2. Secondary Outcome: Change From Baseline to Week 8 in Blepharospasm Disability Index
Description: Blepharospasm Disability Index is a validated 5-point (0-4) scale with six items (e.g., reading, driving a vehicle).
  0 - no impairment, 1 - mild impairment, 2 - moderate impairment, 3 - severe impairment, 4 - not possible due to disease, N/A - Not applicable.
  The total score ranged from 0 (no impairment) to 24 (not possible due to disease). A negative change from baseline indicated improvement.
Time Frame: Baseline to Week 8
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: Points on Scale
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Number analyzed (Participants) | 31 | 33
Points on Scale | -1.3 (3.9) | -0.8 (3.2)

3. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in Total Jankovic Rating Scale (JRS) (Severity and Frequency Measured on a Scale of 0-4)
Description: Jankovic Rating Scale Severity: 0 - None; 1 - Minimal; 2 - Mild; 3 - Moderate; 4 - Severe. Frequency: 0 - None; 1 - Slight increase; 2 - Fluttering duration less than 1 second; 3 - Spasm greater than 1 second and eyes open > 50% of waking time; 4 - Functionally blind. The range of the total score was from 0 (None) to 8 (Severe and Functionally Blind). A negative change from baseline indicated improvement.
Time Frame: Baseline to Week 4 and Week 8
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: Points on Scale
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Number analyzed (Participants) | 31 | 33
Points on Scale
  Change in JRS in Left Eye at Week 4 | -2.3 (1.5) | -1.5 (1.5)
  Change in JRS in Right Eye at Week 4 | -2.2 (1.5) | -1.5 (1.5)
  Change in JRS in Left Eye at Week 8 | -1.9 (1.7) | -1.3 (1.3)
  Change in JRS in Right Eye at Week 8 | -1.8 (1.7) | -1.3 (1.4)

4. Secondary Outcome: Changes From Baseline to Week 4 and Week 8 in Patient Global Assessment (PGA) Score
Description: Subjective satisfaction rating: -4: marked worsening, -3: moderate worsening, -2: marked worsening in symptoms, -1: mild worsening in symptoms, 0: no effect
  +1: mild improvement in symptoms, +2: moderate improvement in symptoms, +3: mild improvement, +4: marked improvement. A positive change from baseline indicated improvement.
Time Frame: Baseline to Week 4 and 8
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: Points on Scale
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Number analyzed (Participants) | 31 | 33
Points on Scale
  Change in PGA at Week 4 | 1.13 (1.86) | 0.52 (2.14)
  Change in PGA at Week 8 | -0.16 (2.37) | 0.19 (1.86)

5. Secondary Outcome: Duration of Action
Description: Median Duration for decision to reinject
Time Frame: Interval between initial injection (Week 0) and final visit (Week 11 through Week 14)
Population: Intention to Treat
Measure: Median (Standard Deviation); unit: Weeks
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Number analyzed (Participants) | 31 | 33
Weeks | 13.1 (2.0) | 13.1 (3.0)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Serious Adverse Events (participants affected / at risk) | 1 | 1
Other Adverse Events (participants affected / at risk) | 21 | 24
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1/31 | 0/33
Carotid Artery Stenosis (Nervous system disorders) | 0/31 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Botulinum Toxin Type A 900kDa | Botulinum Toxin Type A 150kDa
Diplopia (Eye disorders) | 1/31 | 0/33
Dry Eye (Eye disorders) | 0/31 | 1/33
Eye Swelling (Eye disorders) | 0/31 | 1/33
Eyelid oedema (Eye disorders) | 0/31 | 1/33
Lacrimation increased (Eye disorders) | 1/31 | 0/33
Lid Lag (Eye disorders) | 0/31 | 1/33
Sicca Syndrome (Eye disorders) | 0/31 | 2/33
Dry Mouth (Gastrointestinal disorders) | 1/31 | 0/33
Nausea (Gastrointestinal disorders) | 0/31 | 1/33
Salivary hypersecretion (Gastrointestinal disorders) | 0/31 | 1/33
Influenza (Infections and infestations) | 0/31 | 1/33
Periorbital haematoma (Injury, poisoning and procedural complications) | 7/31 | 9/33
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1/31 | 0/33
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1/31 | 0/33
Headache (Nervous system disorders) | 3/31 | 3/33
Mastication Disorder (Nervous system disorders) | 0/31 | 1/33
Paraesthesia (Nervous system disorders) | 0/31 | 1/33
Nervousness (Psychiatric disorders) | 1/31 | 0/33
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/31 | 0/33
Eyelid ptosis (Eye disorders) | 4/31 | 1/33

LIMITATIONS AND CAVEATS:
This was a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less